CLINICAL TRIAL: NCT02785848
Title: Identifying Patient-centered Barriers and Preferred Strategies to Support Self-efficacy for Medication Adherence With Two-way Text Messaging
Brief Title: Identifying Barriers and Strategies to Support Self-efficacy for Medication Adherence With Text Messaging
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Robert M Cronin, MD, MS, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 160750
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asthma and/or Sickle Cell Anemia: The investigators will examine patients with sickle cell disease, asthma, or both who are aged 12-70 years who take daily medications.
  Interventions: Other: Interviews and Surveys

INTERVENTIONS:
Other: Interviews and Surveys — The investigators will perform semi-structured interviews and surveys on this cohort

SUMMARY:
The investigators will explore barriers to improving self-efficacy, or the ability to feel in control of their disease, and medication adherence with text messaging through surveys and interviews with adolescents and adults with SCD cared for at the Vanderbilt Meharry Center of Excellence (VMCE) in Sickle Cell Disease (SCD). The investigators will identify preferences to improve and sustain adherence to daily medication through selection of investigator-proposed or patient-generated text messaging strategies. Finally, the investigators will fill in the literature gaps by describing barriers to self-efficacy and medication adherence among adults with SCD as well as adolescents with SCD who are transitioning to adult care.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving care at the VUMC/Matthew Walker clinic
2. Diagnosed with SCD, asthma, or both
3. Currently taking daily medications for SCD, such as hydroxyurea, asthma, or both
4. Having access to a mobile telephone and/or computer
5. Age 12-70 years

Exclusion Criteria:

1. Unable to perform interviews or surveys

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators will assess barriers to self-efficacy and medication adherence in the adolescents and adults with sickle cell disease (SCD), asthma, or both, who take daily medications such as hydroxyurea, asthma, or both, have access to mobile phones and/or computers and receive care at the VUMC/Matthew Walker clinic.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-05; Primary Completion 2022-05 (Actual); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with barriers to medication adherence | 1 year
  High cost, forgetting, side effects, access to medications

SECONDARY OUTCOMES:
Number of patients that prefer a tailored text messaging technological solution | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cronin, MD, MS, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No